CLINICAL TRIAL: NCT06750107
Title: Testing the Efficacy of Safe South Africa: An Intervention to Prevent HIV Risk and Interpersonal Violence Among Adolescent Boys
Brief Title: Testing the Efficacy of Safe South Africa
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: American University (Other); Medical Research Council, South Africa (Other); Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Caroline Kuo, Associate Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01MH129161 (NIH)
Record Dates: First submitted 2024-12-17; First posted 2024-12-27 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Intervention; Control

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention Safe South Africa (Experimental): This experimental behavioral intervention is designed to (a) lower incidence of sexually transmitted infections (gonorrhea, chlamydia and HIV); and (b) reductions in Intimate Partner Violence (IPV) perpetration frequency and decreased endorsement of IPV supportive attitudes
  Interventions: Behavioral: Safe South Africa
- Control of Standard Care (No Intervention): The control arm will receive standard care. In South Africa, at the time of study planning there are no integrated HIV-IPV interventions that are evidence-based for this age group so the control group will not receive anything, reflective of what would be standard care in this setting.

INTERVENTIONS:
Behavioral: Safe South Africa — The Safe South Africa intervention is a developmentally-tailored intervention for adolescent boys, designed to reduce actual or intended HIV risk behaviors, actual or intended IPV perpetration frequency, and endorsement of IPV supportive attitudes. This intervention comprises 2-hour sessions, held once a week for a total of two weeks. The intervention also includes take-home activities to deepen behavioral engagement with received sessions and to "prime the pump" for up-coming sessions. Part 2 involves behavioral practice, including bystander intervention techniques.
  Arms: Behavioral Intervention Safe South Africa

SUMMARY:
In this study, investigators will examine the efficacy of Safe South Africa, a behavioral intervention that is developmentally- and gender-tailored to prevent human immunodeficiency virus (HIV) and intimate partner violence (IPV) among adolescent boys. South Africa faces some of the highest global rates of HIV and IPV with sustained high incidence of HIV and alarming rates of IPV among adolescents and thus, is an ideal site to advance prevention science to tackle these urgent public health priorities. Testing the efficacy of an integrated intervention to prevent HIV risk behavior and IPV for adolescent boys can support optimal health for young people, their future partners, and society.

DETAILED DESCRIPTION:
Adolescence presents an ideal developmental transition period for an integrated intervention targeting prevention of HIV risk behaviors and intimate partner violence (IPV), including sexual violence. Adolescent boys in particular are at high risk for HIV and perpetration of IPV. Yet, few behavioral interventions integrate HIV-IPV prevention and are tailored for the unique developmental needs of adolescent boys. In this study, investigators build on previous scientific work that demonstrated the acceptability and feasibility of Safe South Africa, an integrated HIV-IPV intervention that uses a developmentally- and gender-tailored approach grounded in social norms theory to prevent adolescent HIV risk behavior and IPV. Investigators will conduct the work in South Africa, a country with the largest HIV epidemic and some of the highest rates of IPV in the world. The investigative team propose the following specific aims: (1) Tailoring Safe South Africa intervention content to address the unique behavioral and social norms data that drives HIV and IPV behaviors among boys in their socioecological environments. (2) Testing the efficacy of the Safe South Africa intervention in preventing HIV/STIs and reducing IPV frequency among N=836 adolescent boys (ages 15- 17), with the scientific team's working hypothesis that the intervention, relative to the usual care condition, will show (a) lower incidence of any STI (including HIV); and (b) reductions in IPV perpetration frequency and decreased endorsement of IPV supportive attitudes. (3) Identifying barriers and facilitators to implementing Safe South Africa within a school setting to provide data for future dissemination (presuming Safe South Africa is efficacious). Investigators will examine processes critical to future dissemination through (a) fidelity data examining adherence to core active components of the standardized intervention manual guiding consistent delivery of the intervention; and (b) qualitative data on the experience during and post-implementation from adolescents and stakeholders using N=20 in-depth interviews with each group.

ELIGIBILITY:
Inclusion Criteria:

* identification as boys
* ages 15-17 years
* enrolled at public high schools in South Africa situated in communities with high rates of HIV and violence

Exclusion Criteria:

* does not have written parental consent
* does not have written assent

Ages: 15 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Identifies as a boy or man
Enrollment: 836 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in incidence of HIV and or Chlamydia and or Gonorrhoeae | 12 months
  Biologically verified Chlamydia trachomatis and/or Neisseria gonorrhoeae and/or HIV are measured as incident infections, defined as the number of participants in the sample who newly acquire HIV and/or Chlamydia and/or Gonorrhoeae as compared to the prior timepoint (this compares 12 month data to baseline). Chlamydia and Gonorrhoeae will be measured using urine sample using an assay (Discharge Multiplex PCR). HIV samples will be captured using a sterile single-person pricking tool is used to create a five dried blood spots card. Samples are tested using a 4th generation assay (Biorad Genscreen ULTRA HIV Ag-Ab assay).
Reduction in acts of intimate partner violence | 12 months
  For those who have engaged in intimate touching, self-reported data on the number of completed acts of forced touching, oral sex, anal sex, and vaginal sex, as well as attempted acts of forced oral, anal, and vaginal sex are collecting using the Sexual Experiences Survey (SES) Short Form Perpetration (SES-SFP) is a survey tool developed by Mary P. Koss (Koss, M. P., Abbey, A., Campbell, R., Cook, S., Norris, J., Testa, M., Ullman, S., West, C., & White, J. (2007). Revising the SES: A Collaborative Process to Improve Assessment of Sexual Aggression and Victimization. Psychology of Women Quarterly, 31(4), 357-370. https://doi.org/10.1111/j.1471-6402.2007.00385.x). The number of participants who have engaged in one or more acts of completed or attempted forced touching are reported at the 12 month timepoint, as compared to prior timepoints.
Lower proportion of those who have reduced endorsement of intimate partner violence supportive attitudes | 12 months
  For those who have engaged in intimate touching, self-reported data on endorsement of IPV supportive attitudes will be measured using the Rape Myth Acceptance Scale. At 12 months, we will compare the proportion of individuals who will lower their Rape Myth Acceptance (RMA) score between baseline and twelve months. The Rape Myth Acceptance Scale is: • Payne DL, Lonsway KA, Fitzgerald LF. Rape myth acceptance: Exploration of its structure and its measurement using the Illinois Rape Myth Acceptance Scale. Journal of Research in Personality 1999;33:27-68.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Kuo, Principal Investigator — American University and Brown University
Locations (1):
- Schools in Cape Town area, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT06750107/Prot_SAP_000.pdf